CLINICAL TRIAL: NCT00430326
Title: A Dose Response Trial to Investigate the Efficacy of Juvista (Avotermin) in the Improvement of Scar Appearance When Applied to Approximated Wound Margins Following Bilateral Varicose Vein Removal.
Brief Title: Juvista (Avotermin) in Scars Following Varicose Vein Removal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Julia Day, Clinical Trial Manager, Renovo
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: RN1001-0042
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Varicose Veins; Cicatrix
MeSH Terms: conditions — Varicose Veins; Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Avotermin

SUMMARY:
This trial is being undertaken to investigate the efficacy and safety of Juvista in the improvement of scar appearance when administered to approximated wound margins following varicose vein surgery. The results from this trial will be used to select doses for investigation in future clinical trials with the compound.

DETAILED DESCRIPTION:
Patients undergoing bilateral removal of the saphenous vein (by ligation and stripping) will be invited to participate in the study. Consenting patients will undergo a detailed screening examination, after which suitability to progress to randomisation to the study will be confirmed.

Suitable screened patients will attend for scheduled surgery of vein removal as normal - this is termed "Day 0" At the time of wound closure, IMP will be administered via intra-dermal injection to each of the incisional groin wounds, and exit wounds.

Each patient will serve as their own control with one leg being administered active IMP (at either a 5, 50, 200 or 500ng/100 ul)of dose solution, whilst the other leg is administered placebo solution. The study is double-blinded, so neither the Investigator nor patient will know which leg wounds receive which treatment.

Further to Day 0, the patients are requested to attend for a further 5 follow up visits (Week 6, Month 3, Month 5, Month 7 & Month 12), where photographs of the scars will be taken, together with spectrophotometry readings to measure colour of the scar. At each visit, the Investigator and patient will rate their opinion of the scar, by global assessment scale & VAS, together with patient completed questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 85 years of age.
* Patients undergoing surgical removal of bilateral varicose veins by ligation and stripping, which will result in clinically similar (i.e. size and location) wounds at the groin and knee.
* Patients who have provided written informed consent.
* Patients with a body mass index between 15 and 35 kg/m2 inclusive.
* Patients with, in the opinion of the Investigator, clinically acceptable results for the laboratory tests specified in the trial protocol (see Protocol Section 6.4.1).
* Female patients of child bearing potential using method(s) of contraception acceptable to the Investigator and who agree to do so from at least the screening visit until one month after administration of the Investigational Medicinal Product.

Exclusion Criteria:

* Patients who have had previous surgical treatment for varicose veins.
* Patients with a history of a bleeding disorder.
* Patients with a chronic or currently active skin disorder which may adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Patients who on direct questioning and/or physical examination, have evidence of any past or present clinically significant medical condition that would impair wound healing.
* Patients who are taking or have taken investigational drugs in the 3 months prior to the screening visit.
* Patients with existing scars within 3cm of the potential trial wounds.
* Patients with diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety, tolerability or efficacy of the Investigational Product.
* Patients with a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Patients who are taking regular, continuous, oral corticosteroid therapy.
* Patients undergoing investigations or changes in management for an existing medical condition.
* Patients who are pregnant or lactating.
* Patients who, in the opinion of the Investigator, are not likely to complete the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Investigator scar assessment | 7 & 12 months
Patient scar assessment | up to 12 months
Independent scar assessment | 7 & 12 months

SECONDARY OUTCOMES:
Local tolerance | ongoing to 12 months
Adverse events | ongoing to12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter McCollum, MB MCh FRCS, Principal Investigator — Hull Royal Infirmary
Locations (21):
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
- P Stradinas Clinical University Hospital, Riga, Latvia
- Lithuania (3):
  - Kaunas 2nd Clinical Hospital, Kaunas
  - Klaipeda Seaman Hospital, Klaipėda
  - Vilnius City University Hospital, Vilnius
- United Kingdom (15):
  - Belfast City Hospital, Belfast
  - Heartlands Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Royal Infirmary, Bristol
  - Derby City General Hospital, Derby
  - Russells Hall Hospital, Dudley
  - Royal Infirmary of Edinburgh, Edinburgh
  - Gloucester Royal Hospital, Gloucester
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - St Georges Hospital, London
  - St Mary's Hospital, London
  - Wythenshawe Hospital, Manchester
  - Freeman Hospital, Newcastle
  - Norfolk & Norwich University Hospital, Norwich

REFERENCES:
- [Derived] McCollum PT, Bush JA, James G, Mason T, O'Kane S, McCollum C, Krievins D, Shiralkar S, Ferguson MW. Randomized phase II clinical trial of avotermin versus placebo for scar improvement. Br J Surg. 2011 Jul;98(7):925-34. doi: 10.1002/bjs.7438. Epub 2011 Mar 29. PMID 21618480